CLINICAL TRIAL: NCT03288831
Title: The Innate Response to and Changes in Intestinal Permeability 4 Hours After a Gluten Challenge in Subjects With Celiac Disease and Non Celiac Gluten Sensitivity
Brief Title: Changes in Intestinal Permeability 4 Hours After Gluten Challenge
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Joseph A. Murray, M.D., Professor of Medicine, Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: IRB 17-003596
Record Dates: First submitted 2017-09-18; First posted 2017-09-20 (Actual); Last update posted 2019-06-07 (Actual); Status verified 2019-06

CONDITIONS: Celiac Disease; Wheat Hypersensitivity; Gluten Sensitivity; Gluten Enteropathy; Immune System and Related Disorders; Duodenal Diseases
Keywords: Randomized, double-blinded, placebo-controlled trial; Oral food challenge
MeSH Terms: conditions — Celiac Disease; Wheat Hypersensitivity; Duodenal Diseases | interventions — Glutens

STUDY DESIGN:
Intervention Model Description: Randomized, double-blinded, placebo-controlled oral gluten challenge
Who Masked: Participant, Care Provider, Investigator
Masking Description: Subjects will be block randomized to either gluten-containing or placebo challenge.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Normal Subjects, Gluten Drink (Active Comparator): Normal subjects will drink a solution containing 6 grams of gluten one time.
  Interventions: Dietary Supplement: Gluten
- Normal Subjects, Placebo Drink (Placebo Comparator): Normal subjects will drink a solution without gluten one time.
  Interventions: Dietary Supplement: Placebo
- Celiac Subjects, Gluten Drink (Active Comparator): Subjects with celiac disease will drink a solution containing 6 grams of gluten one time.
  Interventions: Dietary Supplement: Gluten
- Celiac Subjects, Placebo Drink (Placebo Comparator): Subjects with celiac disease will drink a solution without gluten one time.
  Interventions: Dietary Supplement: Placebo
- Gluten Sensitivity, Gluten Drink (Active Comparator): Subjects with non-celiac gluten sensitivity will drink a solution containing 6 grams of gluten one time.
  Interventions: Dietary Supplement: Gluten
- Gluten Sensitivity, Placebo Drink (Placebo Comparator): Subjects with non-celiac gluten sensitivity will drink a solution without gluten one time.
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Gluten — Six grams of gluten will be mixed with water and Tang flavoring. Subjects will drink the mixture one time.
  Arms: Celiac Subjects, Gluten Drink; Gluten Sensitivity, Gluten Drink; Normal Subjects, Gluten Drink
Dietary Supplement: Placebo — Subjects will drink a mixture of rice water and Tang flavoring one time.
  Arms: Celiac Subjects, Placebo Drink; Gluten Sensitivity, Placebo Drink; Normal Subjects, Placebo Drink

SUMMARY:
This study evaluates why people with celiac disease and non-celiac gluten/wheat sensitivity develop rapid onset symptoms within hours of gluten exposure. Half of subjects will be given gluten and half will not.

DETAILED DESCRIPTION:
When a person with celiac disease is exposed to gluten, their immune system attacks their bowel and causes abdominal pain, bloating, and diarrhea. This process takes 24-72 hours to occur. Some people without celiac disease develop similar symptoms when they eat gluten or wheat. Doctors and scientists do not know what causes this sensitivity to gluten. People with celiac disease and non-celiac gluten sensitivity report symptoms within hours of being exposed to gluten. This study evaluates why this occurs by looking at changes in blood, urine, stool, and the bowel after being given gluten.

ELIGIBILITY:
Inclusion Criteria for subjects with Celiac Disease:

* Biopsy proven celiac disease diagnosed at least 2 years prior to recruitment
* Attest to following a gluten free diet to the best of their ability
* Quiescent symptoms on a gluten free diet
* Negative tissue transglutaminase at time of recruitment (to be collected with baseline blood work)
* A prior endoscopy with small bowel biopsies reviewed by a gastrointestinal pathologist revealing healing

Inclusion Criteria for subjects with Non-Celiac Gluten Sensitivity:

* Meet diagnostic consensus criteria as defined by Ludvigsson et al in "The Oslo definitions for coeliac disease and related terms"
* Attest to following a gluten free diet to the best of their ability
* Quiescent symptoms on a gluten free diet
* Prior negative evaluation for celiac disease (including tissue transglutaminase IgA with total IgA or small bowel biopsies)
* If subjects have had a small bowel biopsies revealing increased intraepithelial lymphocytes (IELs), they will be reviewed as a separate subgroup

Inclusion Criteria for Normal Subjects:

* No gastrointestinal diagnosis (reflux, eosinophilic esophagitis, inflammatory bowel disease, or irritable bowel syndrome)
* No gastrointestinal symptoms (diarrhea, abdominal pain, nausea, vomiting, weight loss)
* No family history of celiac disease
* Will not be required to have a baseline biopsy

Exclusion Criteria:

* Tobacco use
* Symptomatic coronary disease
* Active, severe pulmonary disease
* Baseline oxygen requirement
* Coagulopathy (INR>1.5)
* Mastocytosis
* Active H. pylori infection
* Treated celiac disease with neutrophilia or eosinophilia secondary to infection
* Diabetes (type 1 and type 2)
* Crohn's disease or Ulcerative colitis
* Microscopic colitis
* Dermatitis herpetiformis
* Gastroparesis
* Pregnant women

Subjects exposed to the following medications during their respective time frames will be excluded:

* NSAIDs (24 hours)
* Leukotriene inhibitors (24 hours)
* Mast cell stabilizers (24 hours)
* Benzodiazepines (24 hours)
* H2 blockers (2 days)
* H1 blockers (7 days)
* Steroids (systemic or topically active within gastrointestinal tract) (30 days)
* Topical steroids (14 days)
* Intermittent (up to once weekly) tranquilizer (trazodone, doxepin) use (7 days)
* Chronic tricyclic antidepressant or tranquilizer use (trazodone, doxepin) Use of these medications will also be prohibited during the study duration (AAAAI and AAOA).

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2017-10-10 (Actual); Primary Completion 2018-10-30 (Actual); Study Completion 2018-10-30 (Actual)

PRIMARY OUTCOMES:
Activation of the Mucosal Innate Immune System after Oral Gluten Challenge | 4 hours
  Small bowel biopsies will be assessed for markers of innate immune system activation: presence of granulocytes, granulocyte degranulation, products of degranulation, interleukins and cytokines involved in the innate immune system response, inflammatory mediators.

SECONDARY OUTCOMES:
Changes in Mucosal Permeability after Oral Gluten Challenge | Baseline and up to eight hours after gluten or placebo exposure
  Mucosal permeability will be measure before and after oral gluten or placebo challenge with C13-mannitol lactulose urinary excretion testing. In addition, mucosal permeability will also be measured along the duodenum with a mucosal impedance probe.
Detection of Gluten Peptides in Urine and Stool | Baseline and up to 72 hours after gluten or placebo exposure
  Urine and stool samples will be assessed for the presence of gluten peptides. This will help assess how long these tests are positive after a known gluten exposure.
Rapid Onset Symptom Development after Gluten Exposure | Baseline and up to 72 hours after gluten or placebo exposure
  Subjects will record the symptoms they experience after gluten or placebo exposure. The will complete a simple symptom diary every 30 minutes for the first 2 hours.

CONTACTS AND LOCATIONS:
Overall Officials: Joseph A. Murray, M.D., Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Leffler D, Schuppan D, Pallav K, Najarian R, Goldsmith JD, Hansen J, Kabbani T, Dennis M, Kelly CP. Kinetics of the histological, serological and symptomatic responses to gluten challenge in adults with coeliac disease. Gut. 2013 Jul;62(7):996-1004. doi: 10.1136/gutjnl-2012-302196. Epub 2012 May 22. PMID 22619366
- [Background] Adriaanse MP, Tack GJ, Passos VL, Damoiseaux JG, Schreurs MW, van Wijck K, Riedl RG, Masclee AA, Buurman WA, Mulder CJ, Vreugdenhil AC. Serum I-FABP as marker for enterocyte damage in coeliac disease and its relation to villous atrophy and circulating autoantibodies. Aliment Pharmacol Ther. 2013 Feb;37(4):482-90. doi: 10.1111/apt.12194. Epub 2013 Jan 7. PMID 23289539
- [Background] Anderson RP, van Heel DA, Tye-Din JA, Barnardo M, Salio M, Jewell DP, Hill AV. T cells in peripheral blood after gluten challenge in coeliac disease. Gut. 2005 Sep;54(9):1217-23. doi: 10.1136/gut.2004.059998. PMID 16099789
- [Background] Camarca A, Radano G, Di Mase R, Terrone G, Maurano F, Auricchio S, Troncone R, Greco L, Gianfrani C. Short wheat challenge is a reproducible in-vivo assay to detect immune response to gluten. Clin Exp Immunol. 2012 Aug;169(2):129-36. doi: 10.1111/j.1365-2249.2012.04597.x. PMID 22774987
- [Background] Beitnes AC, Raki M, Brottveit M, Lundin KE, Jahnsen FL, Sollid LM. Rapid accumulation of CD14+CD11c+ dendritic cells in gut mucosa of celiac disease after in vivo gluten challenge. PLoS One. 2012;7(3):e33556. doi: 10.1371/journal.pone.0033556. Epub 2012 Mar 16. PMID 22438948
- [Background] Jansson UH, Kristiansson B, Magnusson P, Larsson L, Albertsson-Wikland K, Bjarnason R. The decrease of IGF-I, IGF-binding protein-3 and bone alkaline phosphatase isoforms during gluten challenge correlates with small intestinal inflammation in children with coeliac disease. Eur J Endocrinol. 2001 Apr;144(4):417-23. doi: 10.1530/eje.0.1440417. PMID 11275953
- [Background] Greco L, D'Adamo G, Truscelli A, Parrilli G, Mayer M, Budillon G. Intestinal permeability after single dose gluten challenge in coeliac disease. Arch Dis Child. 1991 Jul;66(7):870-2. doi: 10.1136/adc.66.7.870. PMID 1863103
- [Background] Horvath K, Nagy L, Horn G, Simon K, Csiszar K, Bodanszky H. Intestinal mast cells and neutrophil chemotactic activity of serum following a single challenge with gluten in celiac children on a gluten-free diet. J Pediatr Gastroenterol Nutr. 1989 Oct;9(3):276-80. doi: 10.1097/00005176-198910000-00003. PMID 2614612
- [Background] Kontakou M, Przemioslo RT, Sturgess RP, Limb GA, Ellis HJ, Day P, Ciclitira PJ. Cytokine mRNA expression in the mucosa of treated coeliac patients after wheat peptide challenge. Gut. 1995 Jul;37(1):52-7. doi: 10.1136/gut.37.1.52. PMID 7672681
- [Background] Strobel S, Busuttil A, Ferguson A. Human intestinal mucosal mast cells: expanded population in untreated coeliac disease. Gut. 1983 Mar;24(3):222-7. doi: 10.1136/gut.24.3.222. PMID 6826106
- [Derived] Cartee AK, Choung RS, King KS, Wang S, Dzuris JL, Anderson RP, Van Dyke CT, Hinson CA, Marietta E, Katzka DA, Nehra V, Grover M, Murray JA. Plasma IL-2 and Symptoms Response after Acute Gluten Exposure in Subjects With Celiac Disease or Nonceliac Gluten Sensitivity. Am J Gastroenterol. 2022 Feb 1;117(2):319-326. doi: 10.14309/ajg.0000000000001565. PMID 34797778
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials